CLINICAL TRIAL: NCT01753401
Title: A Two-part Study Exploring the Efficacy, Safety, and Pharmacodynamics of Acthar in Systemic Lupus Erythematosus Patients With a History of Persistently Active Disease
Brief Title: Acthar for the Treatment of Systemic Lupus Erythematosus (SLE) in Patients With a History of Persistently Active Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QSC01-SLE-01
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2017-08

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Adrenocorticotropic Hormone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 2: Placebo/Acthar (Experimental): Participants receive Placebo in Part 1, but after completion of Week 8 in the double-blind phase, patients who received Placebo may choose to participate in the optional open-label phase where they will receive an Acthar maintenance regimen for 44 weeks. The initial Acthar regimen will be assigned based on the study medication regimen the patient received at the completion of the double-blind phase (Visit 6, Week 8). Acthar regimen during Part 2 may be adjusted based on the Investigator's judgment with the goal of achieving a stable Acthar regimen no later than Week 28. Once the stable Acthar regimen is achieved, the Investigator should consider tapering the steroid regimen to a low daily dose or completely discontinue.
  Interventions: Drug: Acthar; Drug: Placebo; Drug: Steroid Drug
- Period 2: Acthar/Acthar (Experimental): After completion of Week 8 in the double-blind phase, patients who received Acthar may choose to participate in the optional open-label phase where they will receive an Acthar maintenance regimen for 44 weeks. The initial Acthar regimen will be assigned based on the study medication regimen the patient received at the completion of the double-blind phase (Visit 6, Week 8). Acthar regimen may be adjusted based on the Investigator's judgment with the goal of achieving a stable Acthar regimen no later than Week 28. Once the stable Acthar regimen is achieved, the Investigator should consider tapering the steroid regimen to a low daily dose or completely discontinue.
  Interventions: Drug: Acthar; Drug: Steroid Drug
- Period 1: Placebo (Placebo Comparator): Participants receive matching placebo (in 0.5 mL daily or in 1 mL every other day) for 4 weeks. In Weeks 5-8, they will taper the study medication. Participants will continue on their stable steroid regimen during this phase of the study. After completion of Week 8 in the double-blind phase, they may choose to participate in the optional open-label phase. Participants will continue on their stable steroid regimen during this phase of the study.
  Interventions: Drug: Placebo; Drug: Steroid Drug
- Period 1: Acthar (Experimental): Participants receive Acthar (40 units in 0.5 mL daily or 80 units in 1 mL every other day) for 4 weeks. In Weeks 5-8, they will taper the study medication. Participants will continue on their stable steroid regimen during this phase of the study. After completion of Week 8 in the double-blind phase, they may choose to participate in the optional open-label phase. Participants will continue on their stable steroid regimen during this phase of the study.
  Interventions: Drug: Acthar; Drug: Steroid Drug

INTERVENTIONS:
Drug: Acthar — Acthar is given by subcutaneous (SC) injection (shot under the skin), at a dose of 40 units daily or 80 units every other day
  Other Names: H.P. Acthar Gel; Repository Corticotropin Injection
  Arms: Period 1: Acthar; Period 2: Acthar/Acthar; Period 2: Placebo/Acthar
Drug: Placebo — Placebo contains the same inactive ingredients as Acthar, and is given by SC injection
  Other Names: Matching Placebo
  Arms: Period 1: Placebo; Period 2: Placebo/Acthar
Drug: Steroid Drug — The patient's steroid regimen 7.5 to 30 mg/day of prednisone or equivalent, chronic/stable within the 4 weeks prior to screening.
  Other Names: Prednisone or equivalent

SUMMARY:
This Phase 4 study is being performed to examine the effects of Acthar for the indicated use of treatment of SLE. This study will enroll patients with steroid-dependent, persistently active SLE with arthritic and/or cutaneous involvement.

The study will involve two periods: an 8-week double-blind period, to provide placebo-controlled safety, efficacy, and pharmacodynamic data, and an optional open-label period, to examine the prolonged effects of Acthar maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at screening who are able to provide informed consent
* Diagnosis of SLE according to the American College of Rheumatology revised criteria (fulfilled ≥ 4 criteria)
* Active SLE with arthritic and/or cutaneous involvement as demonstrated by a SELENA-SLEDAI score ≥ 2 (clinical manifestation must include rash and/or arthritis)
* Moderate to severe rash and/or arthritis as demonstrated by BILAG score A or B in the mucocutaneous and/or musculoskeletal body systems
* Documented history of autoantibodies to at least one of the following: anti-dsDNA, anti-Smith, or anti-cardiolipin
* Documented history of positive antinuclear antibody (ANA)
* Currently on a stable dose of prednisone (7.5 to 30 mg/day of prednisone or equivalent within the 4 weeks prior to screening). The prednisone regimen must remain stable through the double-blind phase and until the stable Acthar regimen is attained in the open-label phase.

Exclusion Criteria:

* Patients with a recent history (≤ 2 months prior to screening) of starting prednisone (or equivalent) use
* Patients with active nephritis defined as serum creatinine > 2.5 mg/dL or protein creatinine ratio (PCR) > 1.5 g/g, or patients that required hemodialysis within 3 months prior to screening
* Active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident, cerebritis, or CNS vasculitis), requiring therapeutic intervention within 3 months prior to screening
* Type 1 or type 2 diabetes mellitus (history of gestational diabetes mellitus is not an exclusion), or patients currently taking hypoglycemic medication
* History of using certain medications prior to screening:

  1. oral prednisone (or equivalent) > 30 mg/day, any steroid injection, cyclosporine, or non-biologic investigational drug within 3 months prior to screening
  2. intravenous immunoglobulin (IVIg) or plasmapheresis within 4 months prior to screening
  3. cyclophosphamide within 6 months prior to screening; and/or
  4. B-cell targeted therapy, abatacept, or any biologic investigational agent within 12 months prior to screening
* Contraindication per Acthar Prescribing Information: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction

  1. For the purposes of this study, osteoporosis is defined as evidence of vertebral or long bone fracture or vertebral T-score > 2.0
  2. For the purposes of this study, history of peptic ulcer is defined as ≤ 6 months prior to screening
  3. For the purposes of this study, congestive heart failure is defined as New York Heart Association Functional Class III-IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (20):
- United States (20):
  - Mallinckrodt Investigational Site, Jonesboro, Arkansas
  - Mallinckrodt Investigational Site, La Jolla, California
  - Mallinckrodt Investigational Site, La Palma, California
  - Mallinckrodt Investigational Site, Long Beach, California
  - Mallinckrodt Investigational Site, Upland, California
  - Mallinckrodt Investigational Site, Brandon, Florida
  - Mallinckrodt Investigational Site, Clearwater, Florida
  - Mallinckrodt Investigational Site, Miami Lakes, Florida
  - Mallinckrodt Investigational Site, Orlando, Florida
  - Mallinckrodt Investigational Site, Tampa, Florida
  - Mallinckrodt Investigational Site, Granger, Indiana
  - Mallinckrodt Investigational Site, Baton Rouge, Louisiana
  - Mallinckrodt Investigational Site, Lansing, Michigan
  - Mallinckrodt Investigational Site, Brooklyn, New York
  - Mallinckrodt Investigational Site, Great Neck, New York
  - Mallinckrodt Investigational Site, New York, New York
  - Mallinckrodt Investigational Site, Charlotte, North Carolina
  - Mallinckrodt Investigational Site, Hershey, Pennsylvania
  - Mallinckrodt Investigational Site, Wyomissing, Pennsylvania
  - Mallinckrodt Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 enrolled participants were randomized 2:1:2:1 into four treatment groups, to receive Acthar 0.5 mL daily: Placebo 0.5 mL daily: Acthar 1 mL every other day: Placebo 1 mL every other day, during the double-blind period, along with their stable dose of steroids.
Pre-assignment Details: All participants were to receive their stable steroid regimen in addition to the study drug throughout the double-blind period (Period 1). If they completed Period 1, they were invited to participate in an open label period (Period 2). Those who received Placebo went into Placebo/Acthar, and those who received Acthar went into Acthar/Acthar.
Groups:
- Placebo: Participants receive their randomized regimen of placebo during the double-blind period
- Acthar: Participants receive their randomized regimen of Acthar during the double-blind period
- Placebo/Acthar: Participants who receive Placebo in Part 1, but Acthar in Part 2
- Acthar/Acthar: Participants who receive Acthar in both Parts 1 and 2
Period: Double-blind Period (8 Weeks)
Arm/Group | Placebo | Acthar | Placebo/Acthar | Acthar/Acthar
Started | 12 | 26 | 0 (This arm was not included in the double-blind period) | 0 (This arm was not included in the double-blind period)
Modified Intent to Treat (mITT) | 11 | 25 | 0 | 0
Completed | 11 | 22 | 0 | 0
Not Completed | 1 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Open Label Period (44 Weeks)
Arm/Group | Placebo | Acthar | Placebo/Acthar | Acthar/Acthar
Started | 0 (This arm was not included in the open label period) | 0 (This arm was not included in the open label period) | 11 | 22
mITT | 0 | 0 | 11 | 22
Safety Analysis Set | 0 | 0 | 11 | 22
Completed | 0 | 0 | 7 | 13
Not Completed | 0 | 0 | 4 | 9
Not completed — Adverse Event | 0 | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Reason not provided | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received study drug
Groups:
- Placebo: Participants who were randomized to receive Placebo in Period 1
- Acthar: Participants who were randomized to receive Acthar in Period 1
- Total: Total of all reporting groups
Arm/Group | Placebo | Acthar | Total
Number analyzed (Participants) | 11 | 25 | 36
Age, Continuous [Median (Full Range); unit: years] | 39 [27 to 60] | 43 [21 to 60] | 41.5 [21 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 24 | 34
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 5 | 6 | 11
  Black or African American | 6 | 18 | 24
  Other | 0 | 1 | 1
  Hispanic or Latino Ethnicity | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 25 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Meet the Definition of a Responder Within 4 Weeks
Description: Participants are counted as responders based on two SLE indices: the Systemic Lupus Erythematosus Disease Activity Index amended by the SELENA group (SELENA-SLEDAI) and the British Isles Lupus Assessment Group (BILAG) Index.
  * decrease in SELENA-SLEDAI score from 4 to 0 for the arthritis descriptor (highest possible score is 4) and no worsening in other organ systems based on BILAG
  OR
  * decrease in SELENA-SLEDAI score from 2 to 0 for rash (highest possible score is 2) and no worsening in other organ systems based on BILAG
  The BILAG is a transitional index that captures changing severity of clinical manifestations. It has an ordinal scale scoring system by design that produces an overview of disease activity across eight systems. The individual system scores were not intended to be summated into a global score.
Time Frame: within 4 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants who receive Placebo in Period 1
- Acthar: Participants who receive Acthar in Period 1
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
Participants | 3 | 4

2. Secondary Outcome: Number of Participants Who Meet the Definition of a Responder Within 8 Weeks
Description: Participants are counted as responders based on:
  * decrease in SELENA-SLEDAI score from 4 to 0 for arthritis and no worsening in other organ systems based on BILAG
  OR
  * decrease in SELENA-SLEDAI score from 2 to 0 for rash and no worsening in other organ systems based on BILAG
Time Frame: within 8 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
Participants | 3 | 11

3. Secondary Outcome: Score on the SELENA-SLEDAI Within 8 Weeks
Description: SLEDAI was modeled on the basis of clinician global judgment. A participant's SELENA-SLEDAI total score is the sum of all marked SLE-related descriptors on a checklist developed by the SELENA Group (also referred to as hybrid SLEDAI).
  The scores of the descriptors range from 0 to 8. A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
  Rows: Week 2, Week 4, Week 6, Week 8
Time Frame: within 8 weeks
Population: mITT
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
score on a scale
  Week 2: number analyzed (Participants) | 10 | 25
  Week 2 | 10.0 [2 to 12] | 8.0 [2 to 20]
  Week 4: number analyzed (Participants) | 10 | 25
  Week 4 | 9.0 [2 to 12] | 8.0 [4 to 20]
  Week 6 | 8.0 [2 to 12] | 6.0 [0 to 16]
  Week 8 | 9.0 [2 to 16] | 6.0 [0 to 13]

4. Secondary Outcome: BILAG Total Score Within 8 Weeks
Description: The BILAG is a transitional index that captures changing severity of clinical manifestations that produces an overview of disease activity across eight systems.
  The 8 systems are scored on a scale from 0=not present to 4=worse, for the 4 week period before the assessment. The lowest possible score is 0, and the highest possible score is 32. A higher score means the symptoms are worse.
  Rows: Baseline, Week 4, Week 8
Time Frame: within 8 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
score on a scale
  at Baseline | 15.4 (9.55) | 15.7 (5.93)
  at Week 4: number analyzed (Participants) | 10 | 22
  at Week 4 | 10.3 (7.80) | 9.2 (5.36)
  at Week 8: number analyzed (Participants) | 11 | 22
  at Week 8 | 13.5 (8.82) | 6.8 (4.31)

5. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Severity at Baseline
Description: PGA of disease severity on a 100 mm visual analogue scale are categorized to the following: 0 point (none) = 0 mm; 1 point (mild) = >0 - 33.33 mm; 2 points (moderate) = >33.33 - 66.67 mm; and 3 points (severe) = >66.67 - 100 mm. The count of participants in each category is reported.
Time Frame: at Baseline
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
Participants
  None | 0 | 0
  Mild | 1 | 2
  Moderate | 8 | 19
  Severe | 2 | 4
  Missing | 0 | 0

6. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Severity at Week 4
Description: as for outcome 5
Time Frame: at Week 4
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
Participants
  None | 0 | 1
  Mild | 5 | 9
  Moderate | 3 | 11
  Severe | 2 | 1
  Missing | 1 | 3

7. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Severity at Week 8
Description: as for outcome 5
Time Frame: at Week 8
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
Participants
  None | 0 | 2
  Mild | 5 | 12
  Moderate | 3 | 7
  Severe | 3 | 1
  Missing | 0 | 3

8. Secondary Outcome: Number of Tender or Swollen Joints Within 8 Weeks
Description: The doctor counted the number of tender or swollen joints at Baseline, at Week 4, and at Week 8
Time Frame: at Baseline, Week 4, and Week 8 (within 8 weeks)
Population: mITT
Measure: Mean (Standard Deviation); unit: Tender or Swollen Joints
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
Tender or Swollen Joints
  at Baseline | 6.2 (5.40) | 9.6 (6.90)
  at Week 4: number analyzed (Participants) | 10 | 22
  at Week 4 | 3.8 (4.34) | 4.5 (4.94)
  at Week 8: number analyzed (Participants) | 11 | 22
  at Week 8 | 4.0 (6.18) | 3.5 (5.89)

9. Secondary Outcome: Cutaneous Lupus Activity as Measured by the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Within 8 Weeks
Description: The CLASI consists of two scores the first summarizes the activity of the disease while the second is a measure of the damage done by the disease. Activity is scored on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. The CLASI score ranges from 0 to 70, with higher scores indicating more severe skin disease.
  Rows: at Baseline, at Week 4, at Week 8
Time Frame: at Baseline, Week 4 and Week 8 (within 8 weeks)
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
score on a scale
  at Baseline | 6.1 (6.63) | 6.4 (6.33)
  at Week 4: number analyzed (Participants) | 10 | 22
  at Week 4 | 6.3 (4.60) | 4.8 (4.08)
  at Week 8: number analyzed (Participants) | 11 | 22
  at Week 8 | 5.7 (6.87) | 3.7 (4.24)

10. Secondary Outcome: Krupp Fatigue Severity Score (FSS) Within 8 Weeks
Description: The Krupp FSS is a scale to rate disability-related fatigue. Respondents use a scale ranging from 1 ("completely disagree") to 7 ("completely agree") to indicate their agreement with nine statements about fatigue. A visual analogue scale is also included with the scale; respondents are asked to denote the severity of their fatigue over the past 2 weeks by placing a mark on a line extending from "no fatigue" to "fatigue as bad as could be." Higher scores on the scale are indicative of more severe fatigue.
  This validated fatigue severity scale measures impact of fatigue with a 9-item questionnaire, with a 7-point Likert scale for each question. Total score ranges from 0 (best possible outcome) to 63 (worst possible fatigue).
  Rows: at Baseline, at Week 4, at Week 8
Time Frame: at Baseline, Week 4 and Week 8 (within 8 weeks)
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
score on a scale
  at Baseline | 5.374 (0.9840) | 5.648 (1.3091)
  at Week 4: number analyzed (Participants) | 10 | 22
  at Week 4 | 5.379 (1.0697) | 5.298 (1.5401)
  at Week 8: number analyzed (Participants) | 11 | 22
  at Week 8 | 5.404 (1.1699) | 5.152 (1.7858)

11. Secondary Outcome: Mean Score on the Physical Component Scale (PCS) of the Short Form 36 Health Status Questionnaire (SF-36) Within 8 Weeks
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Higher scores indicate improvement.
  Rows: at Baseline, at Week 4, at Week 8
Time Frame: at Baseline, Week 4 and Week 8 (within 8 weeks)
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
score on a scale
  at Baseline | 32.927 (12.3561) | 31.526 (11.7065)
  at Week 4: number analyzed (Participants) | 10 | 22
  at Week 4 | 32.831 (13.5390) | 35.318 (12.5159)
  at Week 8: number analyzed (Participants) | 11 | 22
  at Week 8 | 33.310 (12.9760) | 35.701 (11.8032)

12. Secondary Outcome: Mean Score on the Mental Component Scale (MCS) of the Short Form 36 Health Status Questionnaire (SF-36) Within 8 Weeks
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Higher scores indicate improvement.
Time Frame: at Baseline, Week 4 and Week 8 (within 8 weeks)
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acthar
Number analyzed (Participants) | 11 | 25
score on a scale
  at Baseline | 41.304 (11.8440) | 38.406 (14.6618)
  at Week 4: number analyzed (Participants) | 10 | 22
  at Week 4 | 38.744 (16.8434) | 40.280 (13.0274)
  at Week 8: number analyzed (Participants) | 11 | 22
  at Week 8 | 39.256 (18.4576) | 40.408 (15.8738)

13. Secondary Outcome: Number of Participants Who Meet the Definition of a Responder at Week 52
Description: as for outcome 2
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 7 | 13
Participants | 4 | 3

14. Secondary Outcome: Score on the SELENA-SLEDAI at Week 52
Description: SLEDAI was modeled on the basis of clinician global judgment. A participant's SELENA-SLEDAI total score is the sum of all marked SLE-related descriptors on a checklist developed by the SELENA Group (also referred to as hybrid SLEDAI).
  The scores of the descriptors range from 0 to 8. A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 7 | 13
score on a scale | 3 [0 to 8] | 4 [0 to 10]

15. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Severity at Week 52
Description: as for outcome 5
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 11 | 22
Participants
  None | 0 | 4
  Mild | 7 | 7
  Moderate | 0 | 2
  Severe | 0 | 0
  Missing | 4 | 9

16. Secondary Outcome: Number of Tender or Swollen Joints at Week 52
Description: The doctor counted the number of tender or swollen joints at Week 52.
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Mean (Standard Deviation); unit: Tender or Swollen Joints
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 7 | 13
Tender or Swollen Joints | 1.1 (2.27) | 0.7 (2.21)

17. Secondary Outcome: Cutaneous Lupus Activity as Measured by the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) at Week 52
Description: The CLASI consists of two scores the first summarizes the activity of the disease while the second is a measure of the damage done by the disease. Activity is scored on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. The CLASI score ranges from 0 to 70, with higher scores indicating more severe skin disease.
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 7 | 13
score on a scale | 0.4 (0.79) | 1.3 (1.55)

18. Secondary Outcome: Krupp Fatigue Severity Score (FSS) at Week 52
Description: The Krupp FSS is a scale to rate disability-related fatigue. Respondents use a scale ranging from 1 ("completely disagree") to 7 ("completely agree") to indicate their agreement with nine statements about fatigue. A visual analogue scale is also included with the scale; respondents are asked to denote the severity of their fatigue over the past 2 weeks by placing a mark on a line extending from "no fatigue" to "fatigue as bad as could be." Higher scores on the scale are indicative of more severe fatigue.
  This validated fatigue severity scale measures impact of fatigue with a 9-item questionnaire, with a 7-point Likert scale for each question. Total score ranges from 0 (best possible outcome) to 63 (worst possible fatigue).
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 7 | 13
score on a scale | 4.523 (1.5491) | 4.743 (2.0428)

19. Secondary Outcome: Mean Score on the Physical Component Scale (PCS) of the Short Form 36 Health Status Questionnaire (SF-36) at Week 52
Description: as for outcome 12
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 6 | 13
score on a scale | 43.618 (11.9596) | 39.710 (10.8066)

20. Secondary Outcome: Mean Score on the Mental Component Scale (PCS) of the Short Form 36 Health Status Questionnaire (SF-36) at Week 52
Description: as for outcome 12
Time Frame: at Week 52
Population: mITT with necessary data at Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 6 | 13
score on a scale | 45.272 (12.6597) | 39.700 (16.3027)

21. Secondary Outcome: Number of Participants With a Relapse Within 52 Weeks
Time Frame: within 52 weeks
Population: mITT with necessary data at Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Acthar | Acthar/Acthar
Number analyzed (Participants) | 5 | 19
Participants | 1 | 6

ADVERSE EVENTS:
Time Frame: Period 1: within 8 Weeks of double-blind period, Period 2: within 44 Weeks of open-label period
Description: All treatment-emergent adverse events are listed in the non-serious AE module. Participants are counted only once per term.
Groups:
- Period 1: Placebo: Participants who receive Placebo in Period 1
- Period 1: Acthar: Participants who receive Acthar in Period 1
- Period 2: Placebo/Acthar: Participants who receive Placebo in Period 1, but Acthar in Period 2
- Period 2: Acthar/Acthar: Participants who receive Acthar in both Periods 1 and 2
Arm/Group | Period 1: Placebo | Period 1: Acthar | Period 2: Placebo/Acthar | Period 2: Acthar/Acthar
Serious Adverse Events (participants affected / at risk) | 0/11 | 3/25 | 4/11 | 2/22
Other Adverse Events (participants affected / at risk) | 9/11 | 19/25 | 8/11 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Placebo (N=11) | Period 1: Acthar (N=25) | Period 2: Placebo/Acthar (N=11) | Period 2: Acthar/Acthar (N=22)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Placebo (N=11) | Period 1: Acthar (N=25) | Period 2: Placebo/Acthar (N=11) | Period 2: Acthar/Acthar (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 1
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 2 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1 | 3
Thirst (General disorders) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 2
Blood pressure diastolic increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
False positive investigation result (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 2 | 5 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1
Computerised tomogram thorax abnormal (Investigations) | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1
Percussion test abnormal (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 2 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Non-serious adverse events (AEs) were not tabulated separately for these legacy results, so all treatment emergent adverse events are listed, and serious adverse events might be included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes